CLINICAL TRIAL: NCT01324037
Title: Safety and Feasibility of a Diagnostic Algorithm Combining Clinical Probability, D-dimer Test and Ultrasonography in Suspected Upper Extremity Deep Vein Thrombosis: a Prospective Management Study
Brief Title: Diagnostic Algorithm in Suspected Upper Extremity Deep Vein Thrombosis
Acronym: Armour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Pieter W. Kamphuisen, MD PhD, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL29834.018.09
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Suspected Upper Extremity Deep Vein Thrombosis
Keywords: suspected upper extremity deep vein thrombosis; diagnostic algorithm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clinically suspected upper extremity deep vein thrombosis (Experimental): Patients with suspected upper extremity DVT
  Interventions: Other: diagnostic algorithm

INTERVENTIONS:
Other: diagnostic algorithm — diagnostic algorithm consisting of a clinical decision rule, D-dimer and (serial) ultrasonography

SUMMARY:
Deep vein thrombosis (DVT) of the arm, officially called upper extremity DVT is a rare disorder and accounts for up to 1-4% of all cases of deep vein thrombosis. In case of a thrombosis, there is a blood clot in one of the veins, which should be treated with blood thinners (anticoagulants). The aim of the present study is to see whether it is safe to use a combination of tests for the diagnosis of arm thrombosis. In all patients, we will use a clinical decision rule (clinical judgement) and a laboratory test (D-dimer testing), in most patients also an ultrasound of the arm will be done. The combination of these tests was found to be safe and effective in patients with thrombosis of the legs.

DETAILED DESCRIPTION:
Consecutive patients with clinically suspected upper extremity deep vein thrombosis (UEDVT) are potentially eligible for the study. Patients will be categorized as likely or unlikely to have UEDVT based on a clinical decision rule (CDR). Patients "unlikely" for UEDVT based on the CDR and with normal D-dimer levels will not receive anticoagulant treatment and will be followed-up for 3 months. All patients with a likely CDR or patients with an unlikely CDR combined with elevated D-dimer levels will undergo ultrasonography. In case of an indeterminate ultrasonography result, ultrasonography testing will be repeated 3-5 days later. The same applies for patients with a negative ultrasound and the combination of a high probability and elevated D-dimer levels. Anticoagulants will be withheld in all patients for whom UEDVT will be excluded by the initial diagnostic work-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the emergency department, in and out patient clinic with clinically suspected upper extremity deep vein thrombosis

Exclusion Criteria:

* No informed consent obtained
* Legal age limitation (country specific)
* Use of anticoagulants in therapeutic dosages longer than 24 hours prior to randomisation
* Prior vein thrombosis in the same arm
* Life expectancy < 3 months
* Haemodynamic instability
* Previous participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The cumulative 3-month incidence of objectively confirmed symptomatic venous thromboembolic events including UEDVT and PE in patients with a normal diagnostic work-up. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Willem Kamphuisen, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (18):
- Veterans Affairs Hospital, Washington D.C., District of Columbia, United States
- Austria (2):
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
- University Hospital Leuven, Leuven, Belgium
- University Hospital Dresden, Dresden, Germany
- Italy (5):
  - Ospedali Riuniti, Bergamo
  - University Hospital Bologna, Bologna
  - Hospital D'Annunziata, Chieti
  - University Hospital of Padova, Padua
  - Servizio Sanitario Regionale Emilia - Romagna, Reggio Emilia
- Netherlands (7):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Maxima Medisch Centrum, Eindhoven/Veldhoven
  - University Medical Center Groningen, Groningen
  - Academic Hospital Maastricht, Maastricht
  - Antonius Hospital, Nieuwegein
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Constans J, Salmi LR, Sevestre-Pietri MA, Perusat S, Nguon M, Degeilh M, Labarere J, Gattolliat O, Boulon C, Laroche JP, Le Roux P, Pichot O, Quere I, Conri C, Bosson JL. A clinical prediction score for upper extremity deep venous thrombosis. Thromb Haemost. 2008 Jan;99(1):202-7. doi: 10.1160/TH07-08-0485. PMID 18217155
- [Background] Bernardi E, Pesavento R, Prandoni P. Upper extremity deep venous thrombosis. Semin Thromb Hemost. 2006 Oct;32(7):729-36. doi: 10.1055/s-2006-951458. PMID 17024601
- [Background] Baarslag HJ, van Beek EJ, Koopman MM, Reekers JA. Prospective study of color duplex ultrasonography compared with contrast venography in patients suspected of having deep venous thrombosis of the upper extremities. Ann Intern Med. 2002 Jun 18;136(12):865-72. doi: 10.7326/0003-4819-136-12-200206180-00007. PMID 12069560
- [Background] Di Nisio M, Van Sluis GL, Bossuyt PM, Buller HR, Porreca E, Rutjes AW. Accuracy of diagnostic tests for clinically suspected upper extremity deep vein thrombosis: a systematic review. J Thromb Haemost. 2010 Apr;8(4):684-92. doi: 10.1111/j.1538-7836.2010.03771.x. Epub 2010 Feb 6. PMID 20141579
- [Derived] Kleinjan A, Di Nisio M, Beyer-Westendorf J, Camporese G, Cosmi B, Ghirarduzzi A, Kamphuisen PW, Otten HM, Porreca E, Aggarwal A, Brodmann M, Guglielmi MD, Iotti M, Kaasjager K, Kamvissi V, Lerede T, Marschang P, Meijer K, Palareti G, Rickles FR, Righini M, Rutjes AW, Tonello C, Verhamme P, Werth S, van Wissen S, Buller HR. Safety and feasibility of a diagnostic algorithm combining clinical probability, d-dimer testing, and ultrasonography for suspected upper extremity deep venous thrombosis: a prospective management study. Ann Intern Med. 2014 Apr 1;160(7):451-7. doi: 10.7326/M13-2056. PMID 24687068